CLINICAL TRIAL: NCT04144465
Title: Effect of Noradrenaline Infusuion Versus Phenyephrine Infusion in Improving Tissue Perfusion in HIPEC
Brief Title: Noradrenaline Infusion Versus Phenylephrine Infusion in Improving Serum Lactate Level in HIPEC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, Abdelrhman Alshawadfy, Clinical professor, Suez Canal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: noradrenaline vs phenylephrine
Record Dates: First submitted 2019-10-19; First posted 2019-10-30 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Hyperthermic Intraperitoneal Chemotherapy (HIPEC)
MeSH Terms: interventions — Perfusion; Phenylephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NORADRENALIN (Active Comparator): NORADRENALINE INFUSION
  Interventions: Drug: NORADRENALIN
- PHENYLEPHRINE (Active Comparator): PHENYLEPHRINE INFUSION
  Interventions: Drug: PHENYLEPHRINE

INTERVENTIONS:
Drug: NORADRENALIN — DRUG THAT IS IMPROVING TISSUE AND ORGAN PERFUSION
  Other Names: PERFUSION
  Arms: NORADRENALIN
Drug: PHENYLEPHRINE — DRUG THAT IS IMPROVING TISSUE AND ORGAN PERFUSION
  Arms: PHENYLEPHRINE

SUMMARY:
ABG PARAMETERS ARE CHANGED DURING HIPEC, WE TRIED TO FIND COMPARISON BETWEEN NORADRENALINE AND PHENYLEPHRINE IN OPTIMIZING ABG PARAMETERS THAT REFLECTS ORGAN PERFUSIONS ESPECIALLY SERUM LACTATE

DETAILED DESCRIPTION:
Arterial blood gas testing is considered one of the most important and widely used test in the detection of acidosis, alkalosis, electrolytes disturbance and tissue perfusion. in regard to tissue perfusion serum lactate above 4 mmol/L indicates poor tissue perfusion. serum lactate could be measured at ABG or separately. in this study we will test the effect of both noradrenaline and phenylephrine on lactate level at ABG during the stage of HIPAC in managing abdominal cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* CANCER PATIENTS ENROLLED FOR HIPEC

Exclusion Criteria:

* DRUG SENSITIVITY

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
SERUM LACTATE IN ABG | IMMEDIATELY POSTOPERATIVELY
  LANDMARK FOR TISSUE AND ORGAN PERFUSION

CONTACTS AND LOCATIONS:
Locations (1):
- Suez Canal University, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: No